CLINICAL TRIAL: NCT04656743
Title: Comparison of Genicular Nerve Block and Intraarticular Injection for Postoperative Pain in Knee Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: pain in knee arthroscopy
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Injections, Intra-Articular

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intra-articular injection group (Experimental): will receive ultrasound guided intraarticular injection consisting of 20 mL of 0.25% bupivacaine before surgical procedure. The surgical procedure will be started 30 min after intraarticular injection.
  Interventions: Procedure: intra-articular injection
- genicular nerve block group (Experimental): will receive ultrasound guided genicular nerve block at three nerves, i.e., superomedial, superolateral, and inferomedial genicular nerves consisting of 15 ml bupivacaine 0.25% before surgical procedure. The surgical procedure will be started 30 min after genicular nerve block.
  Interventions: Procedure: genicular nerve block

INTERVENTIONS:
Procedure: intra-articular injection — The injection will be performed under ultrasound guidance by placing the patient's knee in approximately 90° of flexion with the leg hanging off the side of the bed (left). A high-frequency linear transducer ultrasound probe is placed in the superolateral corner of the patella, directed medially toward the patellofemoral joint space. In the extended leg, from anterior to posterior, the right image shows the quadriceps femoris tendon (QF), suprapatellar fat pad (SF), suprapatellar bursa (SB), prefemoral fat pad (PF), and femur (F). When the knee is flexed to 90°, the size of the suprapatellar bursa image is increased. Using an in-plane approach, the needle will be directed into the suprapatellar joint space, and 20 ml of bupivacaine 0.25% will be injected.
  Arms: intra-articular injection group
Procedure: genicular nerve block — The transducer will be first placed parallel to the long bone shaft and moved up or down to identify the epicondyle of the long bone. The genicular arteries will be identified near the periosteal areas, confirmed by color Doppler ultrasound. Accordingly, genicular nerve block target points should be next to each genicular artery. After using color Doppler to confirm the genicular artery, the needle will be inserted in the plane of the ultrasound probe in the long-axis view. a gentle aspiration will be performed and a 2 mL injection volume will be administered.
  Arms: genicular nerve block group

SUMMARY:
This prospective double-blinded randomized study will be conducted to compare ultrasound-guided intra-articular injection and ultrasound-guided genicular nerve block for postoperative analgesia after knee arthroscopy.

DETAILED DESCRIPTION:
Arthroscopic knee surgery has become increasingly popular in modern orthopedics. Post-operative knee pain management has become a challenge to provide early relief and pain-free postoperative care to the patient.

Pain management has become a priority for management as a daycare procedure. Patients operated as a daycare procedure should have minimal postoperative pain which influences the timing of discharge. Pain is due to multifactorial causes such as irritation of free nerve endings of the joint capsule, synovial tissue, anterior fat pad.

Effective pain relief allows the patients to obtain early knee mobilization and optimal rehabilitation and thus improves patient satisfaction.

Postoperative pain after knee arthroscopy is commonly moderate to severe and can affect the patient's activity level and satisfaction.

In an effort to provide safe, effective, and long-lasting post-arthroscopy pain relief, many drug regimens were injected intra-articularly including local anesthetics alone or with additive drugs to prolong and improve the quality of postoperative analgesia.

Genicular nerve block (GNB) and ablation have been used for managing chronic pain from knee osteoarthritis with good success.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for unilateral knee arthroscopy surgery (ligament reconstruction, cartilage procedures, and diagnostic arthroscopic procedures)
* aged between 18 and 50 years
* of both genders,
* have ASA physical status I and II.

Exclusion Criteria:

* Revision knee arthroscopy,
* previous surgery or trauma to the knee,
* drug allergy,
* regular narcotic use,
* renal &/ or hepatic impairments,
* neuromuscular diseases
* and coagulopathy disorders.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
first time of rescue analgesia | postoperative first day
  first time of rescue morphine analgesia

SECONDARY OUTCOMES:
Number of patients received rescue analgesia. | postoperative first day
  number of patients required postoperative rescue morphine analgesis
Total doses of postoperative morphine consumption | postoperative first day
  Total doses of postoperative morphine consumption as rescue analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Tarek Abdel Hay, Tanta, El Gharbyia, Egypt